CLINICAL TRIAL: NCT03982043
Title: Text2Connect, Component 2 of iCHART (Integrated Care to Help At-Risk Teens)
Acronym: T2C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Kaiser Foundation Research Institute (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Tina R Goldstein, Associate Professor of Psychiatry and Psychology, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY18120039; P50MH115838-02 (NIH)
Record Dates: First submitted 2019-06-07; First posted 2019-06-11 (Actual); Results first posted 2022-03-17 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Depression; Suicidal Ideation
MeSH Terms: conditions — Depression; Suicidal Ideation

STUDY DESIGN:
Intervention Model Description: Ultimately, this study design was an open trial after unsuccessful attempts to maintain initial recruitment sites in the study.
  This study initially attempted to use a stepped wedge design, which involves the sequential random rollout of an intervention over 2 time periods. Following a baseline period in which no clusters (= practices) are exposed to the intervention, the crossover is typically in one direction, from control to intervention and continues until both of the clusters have crossed-over to receive the intervention, with observations taken from each cluster and at each time period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Text2Connect (Experimental): Participants receiving Text2Connect (T2C) personalized messages aimed at increasing motivations in at-risk adolescents and their parents. The most salient of the following behavior change techniques will be selected and targeted messaging will be deployed on the participants' phone: psychoeducation, cued mood monitoring, adolescent-parent communication prompts, cognitive bias modification, and cues to action. Intervention material will be tailored to baseline characteristics and T2C will generate reports to providers.
  Interventions: Behavioral: Text2Connect

INTERVENTIONS:
Behavioral: Text2Connect — Text2Connect is a personalized text messaging intervention for patients and parents that targets self-identified barriers to engaging in treatment to increase the likelihood that a depressed or suicidal patient will initiate recommended services.

SUMMARY:
This study proposes to develop and examine a personalized, text-based intervention designed to improve engagement with mental health (MH) treatment.

DETAILED DESCRIPTION:
Text2Connect (T2C) aims to increase perceived susceptibility/severity of depression/suicidality and decrease stigma in at-risk adolescents and their parents. The investigators hypothesize that modification of patient beliefs leads to change talk, thereby increasing the experience of discrepancy which affects motivation for change. These experiences in turn influence decisional balance away from ambivalence toward readiness for change.

Assignment of Interventions:

This study utilized an open trial design. A stepped wedge design was originally proposed and efforts were made to adhere to this study design, however after a year of low recruitment and resultant recruitment sites pulling out the of the study, the overall study design was changed to an open trial. Additional recruitment sites were onboarded to the study and provided with the intervention arm in order to obtain feasibility data on the intervention components of the study. As a result of the change, there are some TAU participants included in this study.

For reference a stepped wedge design involves the sequential random rollout of an intervention over two time periods. Following a baseline period in which no clusters (=practices) are exposed to the intervention, the crossover is typically in one direction, from control to intervention and continues until both of the clusters have crossed-over to receive the intervention, with observations taken from each cluster and at each time period.

This study will pilot Text2Connect in community pediatric and mental health practices using a stepped wedge design (n = 50 adolescents).

Hypothesis: Readiness for mental health care will be greater among adolescents in T2C vs adolescents referred during TAU.

ELIGIBILITY:
Inclusion Criteria:

Youth aged 12-26 yo Own a cell phone with text message capability Biological or adoptive parent is willing to provide informed consent for teen to participate Youth speaks and understands English

* Positive PHQ score or provider determines youth has depressive symptoms based on clinical interaction and refers youth to the study (in cases when PHQ is not available and study staff will complete the PHQ during the screening) OR Provider can refer if they are unclear if symptoms are depressive and PHQ scoring will be used to determine youth's eligibility. OR Screening Wizard screening questionnaire (which includes the PHQ and depressive symptom questions) indicates depression OR provider indicates there is a concern that youth has mood or behavioral problem.
* Referred to mental health care OR screening wizard questionnaire (which indicates if provider makes referral to mental health care)

PHQ-9 scores:

Score of 8 or higher on PHQ-8 -or- Score of 1 or higher on #9 of PHQ-9 suicidality item

Parent inclusion criteria:

Age 18 or older Own a cell phone with text message capability Speaks and understands English Parent of a youth that scores positive on the PHQ-8 or #9 as described above Parent of a youth who has been referred to mental health treatment

Exclusion Criteria:

Non English speaking No parent willing to provide informed consent No cell phone with text messaging capability Is currently experiencing mania or psychosis Evidence of an intellectual or developmental disorder (IDD) Life threatening medical condition that requires immediate treatment Other cognitive or medical condition preventing youth from understanding study and/or participating.

Not referred to mental health care

Parent exclusion criteria:

No cell phone with text messaging capability Child meets exclusion criteria as described above Other cognitive or medical condition preventing parent from understanding study and/or participating.

Ages: 12 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 47 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tina Goldstein, PhD, Principal Investigator — University of Pittsburgh; Brian Suffoletto, MD, Study Director — University of Pittsburgh Medical Center
Locations (4):
- United States (4):
  - CCP Waterdam, McMurray, Pennsylvania
  - Children's Community Pediatrics (CCP-Natrona Heights) of Children's Hospital of Pittsburgh of UPMC, Natrona Heights, Pennsylvania
  - Children's Community Pediatrics (CCP-GIL) of Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - STAR-Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
All requests for study data will follow NIMH's data sharing and data use policies.
  The final completely de-identified dataset(s) will include demographic and clinical data at baseline, and primary and secondary outcomes for all studies, including those funded by the innovation contests. These analytic datasets may also include derived variables with documentation. Our form datasets will include original case report forms, a detailed codebook of variable names, value labels, and programming formats and all study documentation including the protocol and manual of procedures. For descriptive/raw data, study investigators/study staff will upload to NIMH's National Database for Clinical Trials Related to Mental Health Illness (NDCT) on a semi-annual basis all analyzed data being uploaded prior to primary paper publication.
Time Frame: These data will be released to the NDCT soon after each project's "main outcomes" manuscript is accepted for publication.
Access Criteria: In addition to public access to the NDCT, data can also be accessed by contacting ETUDES Center investigators.

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment As Usual (TAU): Participants in the TAU group received a referral for mental health services from their Primary Care Physician (PCP) and did not receive the personalized text messaging intervention.
Period: Overall Study
Arm/Group | Text2Connect | Treatment As Usual (TAU)
Started | 43 | 4
Completed | 43 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Text2Connect | Treatment As Usual (TAU) | Total
Number analyzed (Participants) | 43 | 4 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 28 | 4 | 32
  Between 18 and 65 years | 15 | 0 | 15
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex at Birth: Male | 8 | 1 | 9
  Sex at Birth: Female | 35 | 3 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 41 | 4 | 45
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 33 | 2 | 35
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 43 | 4 | 47

OUTCOME MEASURES:

1. Primary Outcome: Attendance to Treatment
Description: Attendance to the embedded mental health care appointments will be assessed via electronic health record (EHR), as the primary outcome of Text2Connect (T2C)
Time Frame: Week 4 follow up after Baseline
Population: Number of participants who completed the 4-week follow-up questions regarding treatment attendance
Measure: Count of Participants; unit: Participants
Groups:
- Treatment as Usual (TAU): Participants in the treatment as usual (TAU) group received a referral for mental health services from their Primary Care Physician (PCP). Participants in this group did not receive the personalized text messaging intervention, Text2Connect.
Arm/Group | Text2Connect | Treatment as Usual (TAU)
Number analyzed (Participants) | 42 | 4
Participants
  Attended appointment with mental health specialist | 22 | 0
  Did not attend appointment with mental health specialist | 20 | 4

2. Primary Outcome: Attendance to Treatment
Description: as for outcome 1
Time Frame: Week 12 follow up after Baseline
Population: Number of participants who completed 12 week follow-up questions regarding treatment attendance
Measure: Count of Participants; unit: Participants
Arm/Group | Text2Connect | Treatment As Usual (TAU)
Number analyzed (Participants) | 20 | 4
Participants
  Attended appointment with mental health specialist | 8 | 2
  Did not attend appointment with mental health specialist | 12 | 2

3. Secondary Outcome: Number of SMS Messages Answered by Participants
Description: Use of the technical components of T2C will be monitored. Utilization will be measured by the number of participant responses to the automatic T2C SMS messages at the baseline timepoint.
Time Frame: At Baseline phone visit
Population: Number of T2C SMS messages sent to participants between time of screening and baseline assessment
Measure: Count of Units; unit: SMS Sent
Units Other Than Participants: SMS Sent
Arm/Group | Text2Connect
Number analyzed (Participants) | 40
Number analyzed (SMS Sent) | 698
SMS Sent | 621

4. Secondary Outcome: Number of SMS Messages Answered by Participants
Description: Use of the technical components of T2C will be monitored. Utilization will be measured by the number of participant responses to the automatic T2C SMS messages at the 4 week follow-up timepoint.
Time Frame: Week 4 follow up after Baseline
Population: Number of SMS messages sent to participants between baseline and 4 week follow-up assessment.
Measure: Count of Units; unit: SMS Sent
Units Other Than Participants: SMS Sent
Arm/Group | Text2Connect
Number analyzed (Participants) | 24
Number analyzed (SMS Sent) | 744
SMS Sent | 661

5. Secondary Outcome: Number of SMS Messages Answered by Participants
Description: Use of the technical components of T2C will be monitored. Utilization will be measured by the number of participant responses to the automatic T2C SMS messages at the 12 week follow-up timepoint.
Time Frame: Week 12 follow up after Baseline
Population: Number of SMS messages sent to participants between the 4 week and 12 week follow-up assessment.
Measure: Count of Units; unit: SMS Sent
Units Other Than Participants: SMS Sent
Arm/Group | Text2Connect
Number analyzed (Participants) | 9
Number analyzed (SMS Sent) | 366
SMS Sent | 328

6. Secondary Outcome: Service Utilization-Baseline
Description: The Child and Adolescent Service Assessment (CASA) will collect service utilization of all participants to determine the amount of services accessed in each treatment arm. An overall average of the cost of implementing the Text2Connect intervention (including labor, equipment, supplies, facilitates) can be estimated and between the intervention costs and cost of services used from CASA, a comparison will be made and results published. The CASA response data displayed are those who responded positively that they received the service.
Time Frame: At Baseline phone visit
Population: All participants in both treatment and TAU arms completed CASA assessment at Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Text2Connect | Treatment as Usual (TAU)
Number analyzed (Participants) | 43 | 4
Participants
  Use outpatient services | 35 | 1
  Use school services | 30 | 2
  Use ER services | 5 | 0
  Use legal services | 0 | 0
  Use inpatient services | 9 | 0
  Use medications | 30 | 0

7. Secondary Outcome: Service Utilization-Follow Up 4 Weeks
Description: as for outcome 6
Time Frame: Week 4 follow up after Baseline
Population: All participants in both arms completed CASA assessment at 4 week follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | Text2Connect | Treatment as Usual (TAU)
Number analyzed (Participants) | 43 | 4
Participants
  Use outpatient services | 28 | 0
  Use school services | 7 | 1
  Use ER services | 0 | 0
  Use legal services | 0 | 0
  Use inpatient services | 0 | 0
  Use medications | 25 | 0

8. Secondary Outcome: Service Utilization-Follow up 12 Weeks
Description: as for outcome 6
Time Frame: Week 12 follow up after Baseline
Population: 42/43 participants responded to CASA assessment from Text2onnect intervention arm at week 12 and all Treatment As Usual participants completed CASA assessment as week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Text2Connect | Treatment as Usual (TAU)
Number analyzed (Participants) | 42 | 4
Participants
  Use outpatient services | 23 | 0
  Use school services | 6 | 0
  Use ER services | 0 | 0
  Use inpatient services | 0 | 0
  Use legal services | 0 | 0
  Use medications | 26 | 1

9. Secondary Outcome: Usability & Satisfaction
Description: Satisfaction to T2C will be assessed through questions developed by investigators to understand experience with the program. The question investigators have adapted from literature reviews on satisfaction is: "If a friend were in need of a mental health referral, would you recommend Text2Connect to him/her?" The response options include: No, definitely not; No, I don't think so; Yes, I think so; Yes, definitely.
Time Frame: At exit interview either following week 4 study visit or week 12 study visit (depending on when youth attend 1st mental health care appointment)
Population: Of the 43 participants in the T2C intervention group, 40 participants completed the exit interview which included these usability and satisfaction questions.
Measure: Count of Participants; unit: Participants
Arm/Group | Text2Connect
Number analyzed (Participants) | 40
Participants
  No, definitely not | 2
  No, I don't think so | 10
  Yes, I think so | 21
  Yes, definitely | 7

10. Secondary Outcome: Usability & Satisfaction
Description: Satisfaction with the technical components of interventions will be assessed through the certain questions from the Post System Satisfaction and Usability Questionnaire (PSSUQ). The PSSUQ is 19 items with response options ranging from 1 to 7 where 1=strongly disagree and 7=strongly agree. The PSSUQ has sub-scores derived from subsets of the questions which reflect system usefulness, information quality, and interface quality. Questions from sub-domains were chosen to tailor the questioning to this particular intervention. Another question about the need to learn new things before using the app was asked to be rated on a 1-5 scale, with 1= strongly disagree and 5= strongly agree. Two other satisfaction questions included were: "How satisfied are you with the amount of help you received?" The response options were on a scale of 1 (Very dissatisfied) to 4 (Very satisfied). "Have the services you received helped you to deal more effectively with your problems?" The response options were
Time Frame: as for outcome 9
Population: Of the 43 participants in the T2C intervention group, 40 participants participated in the exit interview to answer the PSSUQ.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Text2Connect
Number analyzed (Participants) | 40
score on a scale
  Overall, I am satisfied with how easy it is to use Text2Connect (1 to 7) | 6.1 (1.1)
  The information provided with T2C was clear (1 to 7) | 6.3 (0.9)
  I liked interacting with the T2C program (1 to 7) | 5.1 (1.5)
  I need to learn a lot of things before I could get going with T2C (1 to 5) | 1.4 (1)
  How satisfied were you with the amount of help you received (1 to 4) | 3.1 (0.5)
  Have the services you received helped you to deal more effectively with your problems? (1 to 4) | 2.8 (0.6)

ADVERSE EVENTS:
Time Frame: Over the 1 year and 1 month of data collection for the study, participants were assessed for adverse events at each timepoint (baseline, 4 week follow-up, 12 week follow-up)
Arm/Group | Text2Connect | Treatment As Usual (TAU)
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/4
Other Adverse Events (participants affected / at risk) | 0/43 | 0/4

LIMITATIONS AND CAVEATS:
Limitations included recruiting mostly White females, measuring MH care initiation through adolescent self-report, and not capturing specific MH/substance use diagnoses in addition to depression. Therefore, findings may not be valid in males or racial/ethnic minorities and we were limited in the understanding of severity and breadth of MH care needs.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-02): https://cdn.clinicaltrials.gov/large-docs/43/NCT03982043/Prot_SAP_000.pdf
  • Informed Consent Form (2021-02-02): https://cdn.clinicaltrials.gov/large-docs/43/NCT03982043/ICF_001.pdf